CLINICAL TRIAL: NCT03249779
Title: Electrical Stimulation Via the Scrambler Device as a Treatment for Restless Legs Syndrome/Willis Ekbom Disease
Brief Title: Treatment of RLS/WED Symptoms Through Sensory Counter-stimulation
Acronym: RLS/WED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Melissa Lipford, MD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-005286
Record Dates: First submitted 2016-12-13; First posted 2017-08-15 (Actual); Results first posted 2019-09-04 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Restless Legs Syndrome; Willis-Ekbom Disease
MeSH Terms: conditions — Restless Legs Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Scrambler (Experimental): All participants will receive electrical stimulation applied to the lower extremities using the Scrambler.
  Interventions: Device: Scrambler

INTERVENTIONS:
Device: Scrambler — Scrambler Therapy is a specific form of electrical stimulation which has also been utilized in chronic neurogenic pain11. This modality of therapy differs from TENS in that the goal is to mediate the patient's perception of pain, rather than masking the peripheral pain signal. The results of this modality of treatment may be longer-lasting than TENS, presumably via reduction in central signal generation. Scrambler therapy works through C fibers to retrain the peripheral sensation in the area being treated. Further description of this technology is available at: International Patent PCT/IT2007/000647 and U.S. Patent No. 8,380,317. Literature search does not yield prior studies regarding efficacy of Scrambler therapy in treating RLS

SUMMARY:
To evaluate, in a pilot fashion, efficacy and tolerability of electrical counter-stimulation using the Scrambler device in alleviating uncomfortable sensations and urge to move in patients with restless legs syndrome/Willis Ekbom Disease (RLS/WED).

DETAILED DESCRIPTION:
A total of up to 10 eligible subjects will be recruited who have been diagnosed with chronic RLS/WED (Restless legs syndrome/ Willis Ekbom Disease) in the Mayo Clinic Center for Sleep Medicine. Subjects must experience daily symptoms and must typically be symptomatic during the timeframe in which Scrambler Therapy will be utilized (12-5 PM). Each patient will complete the International Restless Legs Syndrome Rating Scale (IRLS), a validated scale which assesses severity of RLS symptoms16 at baseline (pre-treatment) and before and directly after each session of Scrambler Therapy.

Patients will receive Scrambler Therapy on a daily basis for up to 10 consecutive weekdays. Electrodes will be placed proximal to the area of RLS symptomatology, with gradual downward localization until the entire area of RLS symptoms has been treated. Treatment will initially take place on one leg. Treatments will be administered by a technician trained in using the Scrambler device. A physician or nurse (with familiarity of Scrambler therapy) will be available throughout each treatment session.

Patients will complete questionnaires regarding discomfort or other side effects encountered during or after treatment. Patients will also complete surveys assessing for any changes (benefits or worsening) in RLS symptomatology between treatments.

Patients will be monitored for any adverse events associated with the study procedures. Any reported adverse events will be expediently classified by the study group as to severity level, whether it relates to the treatments in the study protocol, and whether the event was expected or unexpected. This information will allow determination of whether or not the adverse event should be reported as an expedited report or part of the routinely reported outcomes data. All adverse events which meet criteria for expedited reporting will be reported to the institutional IRB as well as external agencies as required.

If there is no evidence of clinical benefit with the first 2-4 patients, then further patients may not be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients age 18 and over diagnosed with RLS/WED by a board certified sleep medicine physician within the Mayo Clinic Center for Sleep Medicine.
* Patients must have moderate to severe symptoms which have been present for ≥ 3 months. Patients must endorse discomfort as part of their typical RLS/WED symptomatology.
* Patients must experience daily symptoms and must experience daily symptoms during afternoon hours (12-5 PM)
* Patients on no medications for RLS/WED, or those who have refractory symptoms despite RLS/WED medications will be enrolled. Patients on alpha-2-delta ligands (pregabalin, gabapentin) will be asked to discontinue these medications two weeks prior to starting treatments and remain off these medications throughout the study protocol.
* Informed consent to participate in this study needs to be obtained

Exclusion Criteria:

* Research authorization not provided
* Patients who are asymptomatic (either by verbal report or completion of severity scale) at time of initiation of Scrambler Therapy treatment
* Patients who have made changes in medication regimen during the 2 weeks prior to study initiation (including initiation of iron supplementation)
* Prior use of Scrambler Therapy
* Pregnant or Nursing Patients
* Patients with implantable drug delivery systems, heart stents, or metal implants (including pacemakers and defibrillators)
* Patients with history of epilepsy or other medical conditions that in the opinion of the investigators should be excluded
* Patients with skin conditions or wounds in or around the area of electrode application (lower extremities)
* Patients treated with alpha-2 delta ligands (gabapentin, pregabalin), who cannot discontinue the medications as above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Lipford, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Scrambler
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Scrambler
Number analyzed (Participants) | 8
Age, Continuous [Mean (Full Range); unit: years] | 71 [51 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in International Restless Legs Syndrome Rating Scale (IRLS)
Description: The International Restless Legs Syndrome Rating Scale (IRLS) questionnaire will be used for this purpose.
  The IRLS is a validated patient-reported outcome measure to accurately assess disease severity of restless legs syndrome. It has questions on the primary features of restless legs syndrome, along with intensity and frequency, associated sleep problems. For this study subjects were asked to answer 10 questions on how often they experienced each symptom, using a score of 0-4, 0 being "None" and 4 being "Very severe." Answers from these questions were combined to provide a total Restless Legs Syndrome score (for a total possible range of 0-40) for each patient at each visit. Lower scores reflected fewer symptoms and higher scores reflected more symptoms.
Time Frame: baseline, 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Scrambler
Number analyzed (Participants) | 8
score on a scale | 19.5 (8.03)
Statistical Analysis 1: Comparison: Scrambler; Test type: Superiority; p = 0.0396, t-test, 2 sided

2. Primary Outcome: Change in International Restless Legs Syndrome Rating Scale (IRLS)
Description: as for outcome 1
Time Frame: baseline, 1 week post treatment (approximately 3 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Scrambler
Number analyzed (Participants) | 8
score on a scale | 20.25 (11.53)
Statistical Analysis 1: Comparison: Scrambler; Test type: Superiority; p = 0.1330, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline through 1 week post treatment, approximately 3 weeks.
Arm/Group | Scrambler
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2016-11-10): https://cdn.clinicaltrials.gov/large-docs/79/NCT03249779/Prot_000.pdf